CLINICAL TRIAL: NCT02592200
Title: A Double Blind Placebo-Controlled Study on the Effect of the Probiotic Lactobacillus Gasseri DSM 27123 on Functional Constipation in Healthy Women - Proof of Concept
Brief Title: Effect of Lactobacillus Gasseri DSM 27123 on Functional Constipation in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0092
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Functional Constipation
Keywords: Female; Constipation; Lactobacillus gasseri DSM 27123; Probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus gasseri (Experimental): Lactobacillus gasseri DSM 27123 capsules, 1×109 CFU (divided in two doses)
  Interventions: Dietary Supplement: Lactobacillus gasseri DSM 27123
- Placebo (Placebo Comparator): Placebo capsules (two doses)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus gasseri DSM 27123 — 109 CFU (divided in two doses) per day for 28 days
  Arms: Lactobacillus gasseri
Dietary Supplement: Placebo — Two doses per day for 28 days
  Arms: Placebo

SUMMARY:
The primary objective is to determine the change in frequency of complete spontaneous bowel movements (CSBMs) after 4 weeks of oral supplementation with Lactobacillus gasseri DSM 27123 in healthy adult women with functional constipation.

DETAILED DESCRIPTION:
Subjects to complete study diaries, number of SBM, CSBM, form of faeces (according to the Bristol Stool Form scale), pain during defecation (according to the visual analogue scale [VAS] 0-100), time spent at each evacuation, episodes of faecal incontinence, number of ingested capsules of investigational product will be recorded daily by the subjects

ELIGIBILITY:
Inclusion Criteria:

The subjects have to meet all of the following criteria to be eligible to enter the study:

1. Willing and able to provide informed consent
2. Women aged 18-49 years at Visit 1
3. BMI ≥18 and ≤29 at Visit 1
4. Suffering of functional constipation as defined by the Rome III criteria for functional constipation
5. Comply with the requirement not to use any other probiotic products from Visit 1 and throughout the study period
6. Not pregnant or breastfeeding
7. Using adequate contraceptive measures
8. Ability to understand and comply with the requirements of the study, as judged by the Investigator

Exclusion Criteria:

1. Hypersensitivity or allergy to the investigational product, to chemically related products or to comparator/placebo
2. Well-known, organic cause of constipation
3. Anorectal pathology
4. Previous gastrointestinal surgery
5. Any alarming symptoms (i.e. rectal bleeding, weight loss, jaundice) as judged by the Investigator
6. Spinal anomalies and injuries
7. Use of antibiotics within 4 weeks prior to Visit 1
8. Use of products containing probiotics more than once a week in the previous 3 weeks
9. Mental or behavioural disorders as judged by the Investigator
10. Food allergy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of complete spontaneous bowel movements (CSBMs) | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change in Stool Consistency (Bristol Stool Form scale) | Baseline, week 1, 2, 3 and 4
  Change in Bristol Stool Form Scale
Change in Patient-Assessment of Constipation Symptoms (PAC-SYM) | Baseline, week 1, 2, 3 and 4 (change from baseline)
  Change in score
Change in Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, week 1, 2, 3 and 4
  Change in Score
Proportion of responders | 4 weeks
  Proportion of responders is defined as subjects showing a mean increase of ≥1 CSBM per week during the treatment period (Day 1 to Day 28) compared to the baseline period (Day-14 to Day -1) or ≥3 CSBMs in the last week of the treatment period (Day 21 to Day 28). The subjects will record time and date of all CSBMs in the study diary.
Number of participants with treatement related adverse events | During the whole study - 4 weeks
  Descriptive
Presence of Lactobacillus gasseri DSM 27123 in faeces | 4 weeks
  qPCR
Need for laxative medication | During the treatment period - 4 weeks
  Time and date of laxative use will be recorded in the study diary by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellström, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- CTC, Akademiska Sjukhuset, Uppsala, Sweden